CLINICAL TRIAL: NCT00004397
Title: Phase I Study of Tin Mesoporphyrin in Patients on Long Term Heme Therapy for Prevention of Acute Attacks of Porphyria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/13187; UTMB-97-117; UTMB-FDR001459
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases | interventions — heme arginate; tin mesoporphyrin

INTERVENTIONS:
Drug: heme arginate
Drug: tin mesoporphyrin

SUMMARY:
OBJECTIVES: I. Evaluate the effectiveness of tin mesoporphyrin in reducing the number of heme infusions needed to prevent acute attacks of porphyria.

II. Evaluate the safety and tolerability of tin mesoporphyrin in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an unblinded study. Patients start a preventive heme regimen and are followed for 6 months prior to tin mesoporphyrin. The frequency of attacks is recorded.

Patients receive tin mesoporphyrin once a week for 6 months. Patients must avoid sunlight during treatment and for 2 months thereafter. The frequency of heme infusions is reduced by half and the frequency of attacks of porphyria is monitored.

Patients are followed for 6 months after last treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Documented acute intermittent porphyria, variegate porphyria, or hereditary coproporphyria causing 6 or more attacks per year Fewer than 2 attacks in the preceding 6 months if already on preventive heme therapy --Prior/Concurrent Therapy-- See Disease Characteristics --Patient Characteristics-- Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Urinary porphobilinogen at least 20 mg/24 hours during acute symptoms Other: Not pregnant Fertile female patients must use effective contraception during and for 6 months prior to study No recurrent symptoms due to another illness No continuous (for longer than 1 month) symptoms of porphyria unless it is in addition to acute exacerbations No acute hemorrhagic disorder such as: Gastrointestinal bleeding Intracerebral hemorrhage No known hypersensitivity to tin mesoporphyrin No known hypersensitivity to any intravenous heme preparation No other condition which may increase risk to patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1998-01; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas